CLINICAL TRIAL: NCT03721614
Title: A Prospective, Active Control, Open-label, Multinational, Randomized Clinical Trial Comparing Single Long BioMimeTM Morph Coronary Stent System vs. Two Overlapping Xience Family Coronary Stent Systems to Evaluate Safety and Performance in Patients With Long de Novo Lesions.
Brief Title: Clinical Study Comparing Single Long BioMimeTM Morph Coronary Stent System vs. Two Overlapping Xience Family Coronary Stent Systems in the Treatment of Patients With Long de Novo Lesions.
Acronym: Morph RCT-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLS/Morph RCT-1
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Study Device :- BioMime™ Morph - Sirolimus Eluting Coronary Stent System Active Control Device :- Xience family Everolimus Coronary Stent Systems
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioMime™ Morph - Sirolimus Eluting Coronary Stent System (Experimental)
  Interventions: Device: BioMime™ Morph - Sirolimus Eluting Coronary Stent System
- Xience family Everolimus Coronary Stent Systems (Active Comparator)
  Interventions: Device: Xience family Everolimus Coronary Stent Systems

INTERVENTIONS:
Device: BioMime™ Morph - Sirolimus Eluting Coronary Stent System — Study Device :- BioMime™ Morph - Sirolimus Eluting Coronary Stent System Approximately 200 patients will be randomly enrolled in a 2:1 ratio [BioMime™ Morph (n=133) vs. XIENCE family (n=67)].
  Arms: BioMime™ Morph - Sirolimus Eluting Coronary Stent System
Device: Xience family Everolimus Coronary Stent Systems — Active Control Device :- Xience family Everolimus Coronary Stent Systems Approximately 200 patients will be randomly enrolled in a 2:1 ratio [BioMime™ Morph (n=133) vs. XIENCE family (n=67)].
  Arms: Xience family Everolimus Coronary Stent Systems

SUMMARY:
A prospective, active control, open-label, multinational, randomized clinical trial comparing single long BioMime™ Morph Coronary Stent System vs. two overlapping Xience family Coronary Stent Systems to evaluate safety and performance in approximately 200 patients with long de novo lesions will be randomly enrolled in a 2:1 ratio [BioMime™ Morph (n=133) vs. XIENCE family (n=67)].

The study population should include patients with symptomatic ischemic heart disease due to de novo lesions (lengths ≥26 mm and ≤56 mm irrespective of number of lesions) in native coronary arteries with a reference vessel diameter of (proximal to distal) 2.75 - 2.25 mm, 3.00 - 2.50 mm and 3.5 - 3.00 mm in patients eligible for Percutaneous Transluminal Coronary Angioplasty (PTCA) and stenting procedures.

All patients must meet all the study inclusion / exclusion criteria before enrolment in the study. All subjects shall accept clinical follow up at 1 month, 6 months, 12 months, 24 months post procedure.

10% of the patients [(2:1) BioMime™ Morph (13) vs. Xience (7)] will be assessed for OCT analysis from pre-designated site(s) and based on availability of OCT console at the site and Patient's consent. [Time Frame: Post-procedure and 6 months (±14 days)]

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least ≥18 years of age.
2. Significant de novo native coronary artery stenosis as part of Ischemic Heart Disease with lesion length of ≥26 mm and ≤56 mm (irrespective of number of lesions) with reference vessel diameter of (Proximal to Distal) 2.75 - 2.25 mm, 3.00 - 2.50 mm and 3.50 - 3.00 mm.
3. Patient with lesion(s), with a visually estimated stenosis of ≥50% and <100% with a TIMI flow of ≥1.
4. Patient must agree not to participate in any other clinical trial for a period of two years following the index procedure. This includes clinical trials of medication and invasive procedures, questionnaire-based studies, or other studies that are non-invasive and do not require medication are allowed.
5. Female patient without childbearing potential who have either undergone surgical sterilization or is post-menopausal.
6. Patient or his/her legally authorized representative (if applicable) agrees to provide written informed consent as approved by respective Ethics Committee and applicable Regulatory Authorities.
7. Patient must agree to undergo all clinical investigations and follow up visits as per protocol.

Exclusion Criteria:

1. Patients with known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, anti-platelet medication specified for use in the study, everolimus and sirolimus, PLLA, PLGA, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
2. Pregnant or nursing patients or those who plan pregnancy in the period up to 2 years following index procedure(Pregnancy should be confirmed based on positive urine pregnancy test as part of screening procedure)
3. An elective surgery planned within 6 months after the procedure that will require discontinuing of DAPT.
4. Patient has a known left ventricular ejection fraction (LVEF) <30% (LVEF may be obtained at the time of the index procedure if the value is unknown and if necessary).
5. Patient has had a known diagnosis of acute myocardial infarction (AMI) preceding the index procedure (CK-MB ≥ 2 times upper limit of normal) and CK-MB/Troponin T/Troponin I values have not returned to within normal limits at the time of procedure.
6. Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or within one year after the index procedure.
7. Patient has undergone heart transplant or any other organ transplant or planned to undergo any organ transplant.
8. Patient is receiving immunosuppressant therapy and/or has known immunosuppressive or autoimmune disease.
9. Patient with active bleeding disorders.
10. Patient has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3, a White Blood Cell count of <3,000 cells/mm3 or documented or suspected liver disease (including laboratory evidence of Hepatitis B and C)
11. Known renal insufficiency (e.g., estimated Glomerular Filtration rate <60 ml/kg/m² or Serum Creatinine level of > 2.0 mg/dL, or patient on dialysis).
12. Patient has had a Cerebrovascular Accident (CVA) or Transient Ischemic Neurological Attack (TIA) within the past 6 months.
13. Patient belonging to a vulnerable population (per Investigator's judgment, e.g., subordinate hospital staff or Sponsor staff).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-22 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 6 months (±14 days)
  Target lesion failure is defined as a composite of cardiac death, myocardial infarction attributed to target vessel or Ischemia-driven target lesion revascularization.

SECONDARY OUTCOMES:
Target Lesion Failure | 1 month (± 7 days), 12 months (±1 month) and 24 months (±1 month)
  Target lesion failure is defined as a composite of cardiac death, myocardial infarction attributed to target vessel or ischemia-driven target lesion revascularization.
MACE | 1 month (± 7 days), 6 months (±14 days), 12 months (±1 month) and 24 months (±1 month)
  Major adverse cardiac event is defined as a composite of cardiac death, myocardial infarction attributed to the target vessel or Ischemia-driven Target Lesion Revascularization (ID-TLR).
Stent Thrombosis Rate (As per Academic Research Consortium) | 1 month (± 7 days), 6 months (±14 days), 12 months (±1 month) and 24 months (±1 month)
  Stent thrombosis is defined by ARC criteria as definite (angiographic confirmation with at least one of the following: acute onset of ischemic symptoms at rest, new ischemic changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers, probable (any unexplained death within the first 30 days), and possible (any unexplained death from 30 days after intracoronary stenting until end of trial follow-up). Stent thrombosis is categorized as acute (0-24 hours post stent implantation), Subacute (>24 hours to 30 days post stent implantation), late (>30 days to 1 year post stent implantation), or very late (>1 year post stent implantation).
Ischemia-driven Target Vessel Revascularization (ID-TVR) | 1 month (± 7 days), 6 months (±14 days), 12 months (±1 month) and 24 months (±1 month)
  Ischemia-driven Target Vessel Revascularization is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.

OTHER OUTCOMES:
Clinical Success | Within 48 hours after the index procedure or at hospital discharge, whichever is sooner
  On a per patient basis, technical success without complications within 48 hours after the index procedure or at hospital discharge, whichever is sooner.
User ratings on technical properties | Baseline]
  User's satisfaction Rating on a scale of 0 - 5 on the parameters of the coronary listed below:
  a) Flexibility b) Pushability c) Trackability d) Crossability e) Inflation time f) Deflation time g) Ease of removal h) Radiopaque marker visibility (Where 0=very poor comfort, 1=poor comfort, 2=below average, 3=average, 4=good and 5=excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ertugrul Okuyan, Principal Investigator — Bagcilar Egitim ve Arastirma Hastanesi; Dr. Omer Kozan, Principal Investigator — Siyami Ersek Gogus Kalp ve Damar Cerrahisi Egitim ve Arastirma Hastanesi; Dr. Jan - Peter V Kuijk, Principal Investigator — St. Antonius Hospital; Dr. Jakub Podolec, Principal Investigator — Krakowski Szpital Specjalistyczny im. Jana Pawla II; Dr. Andrzej Ochala, Principal Investigator — Zaklad Kardiologii Inwazyjnej; Dr. Oleg Polonetsky, Principal Investigator — National Scientific and Practical Centre - Cardiology; Dr. Orazbek Sakhov, Principal Investigator — City Heart Center